CLINICAL TRIAL: NCT03388229
Title: Association Between Dietary Pattern and Glycemic Control Among Type 2 Diabetes Patients in the United Arab Emirates: A Retrospective Cross-sectional Study
Brief Title: Association Between Dietary Pattern and Glycemic Control Among Type 2 Diabetes Patients in the Unites Arab Emirates
Status: Completed | Type: Observational
Sponsor: Rashid Centre for Diabetes and Research (Other)
Responsible Party: Principal Investigator, Dr.Amena Sadiya, Team Leader-Lifestyle Clinic, Rashid Centre for Diabetes and Research
Other Study IDs: DietpatternUAE
Record Dates: First submitted 2017-12-18; First posted 2018-01-02 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Dietary Habits
Keywords: Dietary pattern; glycemic control; type 2 diabetes; UAE
MeSH Terms: conditions — Feeding Behavior; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: not an intervention — it was observation not intervention

SUMMARY:
Poor glycemic control in patients with Type 2 Diabetes (T2D) is due to multiple factors and suboptimal dietary pattern is one of them .Assessing eating/dietary patterns (combinations of different foods or food groups) among individuals with diabetes may be beneficial in understanding the focus areas of dietary modification among the Emirati community and further developing dietary interventions for management of T2D. Only a few observational studies are reported in this region exploring the eating practices, although none to the investigators knowledge described the frequency of consumption of food groups in the T2D patients in the United Arab Emirates(UAE). Hence, in this study the investigators aim to describe the trends in frequency of consumption of food groups and analyze the association of frequency of food item consumption and glycemic control among the T2D UAE patients.

This retrospective cross sectional study will include the data from Hospital information system of 800+ T2D patients to describe the trends in frequency of consumption of food groups and analyze the possible association of frequency of food group/item consumption and glycemic control.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) burden is not only increasing globally but also in the middle east region. Dietary intake plays a crucial role in ameliorating glycemia and other risk factors ,The aim of this study is to describe the trends in frequency of consumption of food groups and possible association with glycemic control among theT2D UAE patients.

This retrospective cross-sectional study was conducted among 800+ T2D diabetic aged ≥ 18 years, attending Rashid Centre for Diabetes and Research(RCDR) Centre located in UAE during January 2011 until January 2015. The dietary data will be collected from hospital records generated by dietitians after an interview based consultation using a structured pre-tested questionnaire. Multiple regression techniques will be used for model building, to determine the separate contribution of known confounders and food items with high carbohydrate and glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* UAE nationals,
* both males and females.
* Age between ≥ 18years

Exclusion Criteria:

* Patients underwent bariatric surgery
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending Rashid Centre for Diabetes and Research care centre located in Ajman, UAE during January 2011 until January 2015.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
association between frequency of food group/item consumption and HbA1c among T2D patients | January 2011 until January 2015
  to develop a regression model of association between frequency of food consumption and poor glycemic control (HbA1c<7%)

SECONDARY OUTCOMES:
To measure the percentage of frequency of consumption of food groups among T2D patients , | January 2011 until January 2015
  assess the food frequency consumption of food groups and food items

CONTACTS AND LOCATIONS:
Locations (1):
- Rashid Centre for Diabetes and Research, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sadiya A, Mnla R. Impact of food pattern on glycemic control among type 2 diabetic patients: a cross-sectional study in the United Arab Emirates. Diabetes Metab Syndr Obes. 2019 Jul 16;12:1143-1150. doi: 10.2147/DMSO.S209320. eCollection 2019. PMID 31406470